CLINICAL TRIAL: NCT01086449
Title: Safety and Immunogenicity of GSK Biologicals' Herpes Zoster Vaccine 1437173A in Healthy Ethnic Japanese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113819
Record Dates: First submitted 2010-03-04; First posted 2010-03-15 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Herpes Zoster
Keywords: safety; Japanese; Herpes Zoster; immunogenicity; Herpes Zoster in healthy ethnic Japanese adults; Vaccine
MeSH Terms: conditions — Herpes Zoster

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: Herpes Zoster Vaccine GSK 1437173A

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK 1437173A — Investigational vaccine (GSK 1437173A) administered intramuscularly.

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of GSK Biologicals' candidate Herpes Zoster (HZ) vaccine in healthy ethnic Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* A male or female between, and including, 18 and 30 years of age at the time of the first vaccination for inclusion in the young adults cohort or aged between, and including, 50 and 69 years of age at the time of the first vaccination for inclusion in the older adults cohort.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Japanese ethnic origin (defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese).
* Female subjects of non-childbearing potential may be enrolled in the study.

  - Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.
* Male subjects may be enrolled in the study, if the subject:

  * has agreed to practice adequate contraception (until 2 months after completion of the vaccination series).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine/product, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine/product dose. For corticosteroids, this will mean prednisone >= 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Concurrent or planned participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Immunosuppression resulting from haematopoietic stem cell transplantation, AIDS or symptomatic HIV infection.
* Previous vaccination against HZ (either a registered product or an investigational product through participation in a HZ vaccine study).
* History of HZ.
* History of any allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Receipt of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Receipt of any other immunisations within one month before the first study vaccination (2 weeks in the case of inactivated influenza vaccines or other non-replicating immunisation products [e.g., tetanus and reduced dose diphtheria toxoid (dT) vaccine, pneumococcal vaccine, hepatitis A vaccine, hepatitis B vaccine]), or scheduled within 30 days after study vaccination.
* Acute disease and/or fever at the time of enrolment.
* Fever is defined as temperature >= 37.5°C (99.5°F) on axillary setting;
* Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions (if of child bearing potential).
* Male planning to father a child or planning to discontinue contraceptive precautions.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2010-06-25 (Actual); Study Completion 2010-11-25 (Actual)

PRIMARY OUTCOMES:
Solicited local and general symptoms | Day 0-6 after each vaccination
Unsolicited adverse events | Day 0 -29
Serious adverse events | From dose 1 up to the end of the study
Occurrence of pre-defined adverse events | From dose 1 up to study end
Haematological and biochemical parameters | Months 0, 1 and 3

SECONDARY OUTCOMES:
Antigen and virus-specific antibody concentrations at protocol-defined time points | Months 0, 1 and 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lal H, Zahaf T, Heineman TC. Safety and immunogenicity of an AS01-adjuvanted varicella zoster virus subunit candidate vaccine (HZ/su): a phase-I, open-label study in Japanese adults. Hum Vaccin Immunother. 2013 Jul;9(7):1425-9. doi: 10.4161/hv.24269. Epub 2013 Apr 12. PMID 23584252
- See also: Results for study 113819 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/113819?search=study&b%22b''%22#rs
- Available data/document: Informed Consent Form: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113819 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register